CLINICAL TRIAL: NCT06056973
Title: A Multicenter, Randomized, Controlled Clinical Trial of Jinghua Weikang Capsule for Maintenance Treatment of Reflux Esophagitis
Brief Title: Jinghua Weikang Capsule in the Treatment of Reflux Esophagitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, zhijun Duan, A multicenter, randomized, controlled clinical trial of Jinghua Weikang Capsule for maintenance treatment of reflux esophagitis, The First Affiliated Hospital of Dalian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PJ-KS-KY-2023-337(X)
Record Dates: First submitted 2023-09-18; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Reflux Esophagitis
MeSH Terms: conditions — Esophagitis, Peptic | interventions — jinghua weikang

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trials group (Experimental): PPI treatment for 8 weeks, ( d1-d56 ), Jinghua weikang capsules 2 tid, 28 days of treatment.
  Interventions: Drug: jinghua weikang capsule
- Control group (Active Comparator): Control group ( 130 cases ) : PPI treatment for 8 weeks, ( d1-d56 ), PPI treatment for 28 days.
  Interventions: Drug: jinghua weikang capsule

INTERVENTIONS:
Drug: jinghua weikang capsule — Oral Jinghua Weikang Capsule, two capsules each time, three times a day

SUMMARY:
Reflux esophagitis is a common clinical disease ; pPI or potassium competitive acid blocker ( P-CAB ) is the first choice for the treatment of reflux esophagitis. However, patients with recurrent symptoms and severe esophagitis ( Los Angeles grade C and D ) after long-term use of PPI or P-CAB usually need long-term maintenance treatment. Attention should be paid to the possible adverse reactions of long-term acid suppression therapy and the interaction between drugs. The main efficacy of Jinghua Weikang capsules is regulating qi and dispersing cold, clearing heat and removing blood stasis. Applicable to cold and heat syndrome, qi stagnation and blood stasis caused by epigastric distension, pain, belching, acid reflux, noisy, bitter taste ; duodenal ulcer see the above syndrome. In the early stage, a series of studies were carried out on Jinghua Weikang Capsule, which confirmed that Jinghua Weikang Capsule showed the effect of acid inhibition and symptom relief in the treatment of reflux esophagitis, and had a synergistic effect when combined with western medicine. However, Jinghua Weikang Capsule still lacks sufficient evidence to support the reduction of the recurrence rate of reflux esophagitis. Therefore, we carried out this experiment to explore the clinical efficacy of Jinghua Weikang Capsule in the maintenance treatment of reflux esophagitis, so as to reduce the recurrence rate of reflux esophagitis and relieve symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent.
* Men and women are not limited
* Age 18-70 years old
* Have been diagnosed as reflux esophagitis, and had recurrence after standard treatment ;
* Upper gastrointestinal endoscopy ( within 1 year ) had reflux esophagitis. In order to facilitate the observation of treatment time and effect, this project selected Los Angeles classification as reflux esophagitis A and B grade.
* GERD questionnaire reached 8 points in patients with
* Have appropriate organs and hematopoietic function, according to the following laboratory tests ( within 1 year ) Neutrophil count ( NEUT # ) ≥ 1.5 × 109 / L ; platelet count ≥ 75 × 109 / L ; hemoglobin ≥ 90g / L ; serum total bilirubin ( TBIL ) ≤ 2 times ULN ; alanine aminotransferase ( ALT ), aspartate aminotransferase ( AST ) ≤ 5 times ULN ; serum albumin ≥ 29 g / L ; serum creatinine ≤ 1.5 times the upper limit of normal ( ULN ) or creatinine clearance rate ≥ 50 mL / min.
* Normal electrocardiogram

Exclusion Criteria:

* Patients who received antibiotics, bismuth, H2RA and PPI treatment within two weeks before the first medication ;
* pregnant or lactating women ;
* patients with moderate or above depression and mental disorders ;
* Patients with dysphagia and peptic ulcer such as achalasia, esophageal cancer ;
* patients with severe liver disease, heart disease, kidney disease, malignant tumor and alcohol dependence ;
* Those who are allergic to the drugs used in this study ;
* Patients who participated in other clinical studies within 3 months ;
* Patients who can not correctly express their complaints and have poor compliance ;
* There are other serious physical or mental illnesses or laboratory abnormalities that may increase the risk of participating in the study, or interfere with the results of the study, and subjects who the researchers believe are otherwise unfit to participate in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Reduce the recurrence rate of R reflux esophagitis and relieve symptoms | 9 months
  To explore the clinical effect of Jinghua Weikang Capsule on the maintenance treatment of reflux esophagitis, in order to reduce the recurrence rate of reflux esophagitis and relieve symptoms.